CLINICAL TRIAL: NCT00900471
Title: Advanced Tumor Bank Project
Brief Title: Collection and Storage of Tissue Samples From Patients Undergoing Surgery For Suspected Solid Tumors
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: BG04-104; P30CA012197 (NIH); CCCWFU-01403; CCCWFU 01403 (Other: WFCCC)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Solid Tumors Tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: biologic sample preservation procedure
Other: medical chart review

SUMMARY:
RATIONALE: Collecting and storing samples of tissue or blood from patients with cancer for study in the laboratory may help the study of cancer in the future

PURPOSE: This research study is collecting and storing blood and tissue samples from patients with suspected solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To provide a tissue and cell repository to be used by Wake Forest University Comprehensive Cancer Center (WFUCCC) investigators.
* To provide specialized research pathology services to these investigators.

OUTLINE: Tumor and normal tissue in the resected specimen (when possible) are harvested and collected from patients undergoing planned surgery or biopsy. Additionally, any normal tissue and/or fluid removed in the course of the operation (e.g., cerebrospinal fluid during brain tumor resection) may also be stored for use in analyzing changes from normal tissue to cancerous tissue. Specimens are rapidly frozen in liquid nitrogen to preserve the mRNA, proteins, lipids, and DNA in the samples for future analysis. Tissue is stored for research projects on tumors and treatment of cancer patients. Research may involve analysis of the genetic makeup of the tumor tissue. Genes may be cloned and living cells cultured from the stored tissue. Blood is also collected during surgery. Samples are maintained and cataloged for future retrieval.

Information about medical history is collected from patient medical records. This information includes the following: medical diagnosis; specific information about treatment; other medical conditions; medical data (i.e., laboratory test results, tumor measurements, CT scans, MRI scans, x-rays, and pathology results); side effects experienced and treatment for side effects; long-term information about general health status and the status of disease; data that may be related to tissue and/or blood samples collected; and identifying numbers or codes (i.e., social security number and medical record number).

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected solid tumor AND scheduled for surgical resection and/or biopsy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those with a clinically suspected solid tumor and scheduled for surgical resection and/or biopsy
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2004-04-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Tissue and cell repository for Wake Forest University Comprehensive Cancer Center investigators | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Edward A. Levine, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States